CLINICAL TRIAL: NCT06577610
Title: The Impact of a Colonoscopy Monitoring Program on Endoscopists' Performance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Su Jin Chung, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2406-162-1549
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Adenoma Colon Polyp; Sessile Serrated Adenoma
Keywords: adenoma; Sessile Serrated Adenoma; colonoscopy
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Feedback group (Experimental): The feedback group will be notified of the colonoscopy performances.
  Interventions: Behavioral: Feedback from colonoscopy monitoring program
- Control group (No Intervention): The control group will not be notified of the colonoscopy performances.

INTERVENTIONS:
Behavioral: Feedback from colonoscopy monitoring program — Adenoma detection rate feedback from colonoscopy monitoring programs
  Arms: Feedback group

SUMMARY:
The goal of this clinical trial is to learn if colonoscopy monitoring program works to adenoma detection rate in endoscopists. It will also learn about the impact on sessile serrated lesion detection rate, adenomas per colonoscopy, sessile serrated lesions per colonoscopy, advanced adenoma detection rate. The main questions it aims to answer are:

Does colonoscopy monitoring program effect on adenoma detection rate in endoscopists?

Participants will:

Receive result of colonoscopy monitoring program or not every 3 months for 1 year

ELIGIBILITY:
Inclusion Criteria:

* Endoscopists with at least 1 year of colonoscopy experience

Exclusion Criteria:

* Endoscopists with less than 1 year of colonoscopy experience

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
adenoma detection rate | 1 year
  the percentage of patients with at least one histologically proven adenoma

SECONDARY OUTCOMES:
sessile serrated lesion detection rate | 1 year
  the percentage of patients with at least one histologically proven sessile serrated lesion
adenomas per colonoscopy | 1 year
  the number of detected adenomas divided by the total number of screening colonoscopies
sessile serrated lesions per colonoscopy | 1 year
  the number of detected sessile serrated lesions divided by the total number of screening colonoscopies
advanced adenoma detection rate | 1 year
  the percentage of patients with at least one histologically proven advanced adenoma

IPD SHARING:
Plan to Share IPD: No